CLINICAL TRIAL: NCT02371252
Title: Randomized Trial Comparing Efficacy and Safety of Brand Versus Generic Alendronate for Osteoporosis Treatment
Brief Title: Efficacy and Safety of Brand Versus Generic Alendronate for Osteoporosis Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 150/2557(EC3)
Record Dates: First submitted 2014-09-07; First posted 2015-02-25 (Estimated); Results first posted 2021-09-29 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Bisphosphonates; Alendronate; Bone mineral density; Bone markers
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Original alendronate (Fosamax) (No Intervention): The patients will be given the brand alendronate (Fosamax®) (70 mg) 1 tablet once a week orally for 1 year after enrollment. In addition, calcium and vitamin D supplementation will be given to all patients.
- Generic alendronate (Bonmax) (Active Comparator): The patients will be given the generic alendronate (Bonmax®) (70 mg) 1 tablet once a week orally for 1 year after enrollment. In addition, calcium and vitamin D supplementation will be given to all patients.
  Interventions: Drug: Generic alendronate

INTERVENTIONS:
Drug: Generic alendronate — The patients will be given the generic alendronate 1 tablet per week for approximately 1 year after enrollment.
  Other Names: Bonmax
  Arms: Generic alendronate (Bonmax)

SUMMARY:
Osteoporosis is a common disease defined as a decrease in bone mass and strength which increases risk of fragility fractures. This disorder may affecting health in many adults which causing disability, morbidity, and mortality. Current first-line medical therapy is bisphosphonates which alendronate is one of the most widely used. However, expenditure on medicines is one of the major problem of inadequate access to treatment.

The investigators hypothesized that generic alendronate will have the same clinical efficacy as the brand formulation. Therefore, the result of this study is extremely crucial. If adequate efficacy of generic alendronate could be established and if it affords the same safety profile as those of brand alendronate, the use of generic alendronate could then be recommended.

DETAILED DESCRIPTION:
Osteoporosis is a common disease which estimated that over 200 million people worldwide are suffered. The prevalence is continuing to escalate with the increasingly elderly population. The risk of fragility fractures in elder over age 50 is approximately 50% in women and 20% in men.

Current first-line medical therapy is bisphosphonates which alendronate is one of the most widely used. However, expenditure on medicines is one of the major problem of inadequate access to treatment. Generally, insurances and health care providers prefer physicians to prescribe generic instead of brand drug, due to its lower costs. However, clinical information on bone mineral density (BMD), fracture reduction and side effects with new generic alendronate is limited.

The objective of this study is to evaluate the efficacy and safety of a new generic alendronate (Bonmax®) comparing to brand alendronate (Fosamax®). The efficacy of generic alendronate will be determined by measuring the percent changes of bone mineral densities at lumbar spine and total hip after 1 year of treatment and then comparing to those changes in the brand alendronate group.

ELIGIBILITY:
Inclusion Criteria: patients who are postmenopausal women or men who aged older than 50 years and meet the indications for osteoporosis treatment according to the Thai Osteoporosis Foundation's 2010 treatment guidelines.

* History of spinal or hip fractures with low energy trauma.
* BMD by Dual energy X-ray absorptiometry (DXA) scan with T-score ≤ -2.5 at the femoral neck, total hip, or L1-L4 spine.
* BMD by DXA scan with T-score between -1 and -2.5 at the femoral neck, total hip, or L1-L4 spine and a 10-year hip fracture probability ≥ 3% or a 10-year major osteoporosis-related fracture probability ≥ 20% based on Fracture risk assessment tool (FRAX)

Exclusion Criteria:

* Patients who have contraindications to use bisphosphonates e.g. gastroesophageal reflux disease or drug allergy to bisphosphonates
* Patients with an abnormality of serum calcium levels (more than 10.2 mg/dl or less than 8.7 mg/dl)
* Patients with estimated glomerular filtration rate less than 30 mL/min/1.73 m2
* Patients with metabolic bone diseases such as Paget's disease, hyperparathyroidism, etc.
* Patients who were received anti-osteoporotic drugs during the past 1 year.
* Patients who currently taking steroids, hormone replacement therapy, or selective estrogen receptor modulators (SERMs) within 1 year.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aasis Unnanuntana, MD, Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Unnanuntana A, Jarusriwanna A, Songcharoen P. Randomized clinical trial comparing efficacy and safety of brand versus generic alendronate (Bonmax(R)) for osteoporosis treatment. PLoS One. 2017 Jul 5;12(7):e0180325. doi: 10.1371/journal.pone.0180325. eCollection 2017. PMID 28678853

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Original Alendronate (Fosamax) | Generic Alendronate (Bonmax)
Started | 70 | 70
Completed | 70 | 70
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Original Alendronate (Fosamax) | Generic Alendronate (Bonmax) | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.7 (9.7) | 73.7 (7.2) | 73.7 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 61 | 127
  Male | 4 | 9 | 13

OUTCOME MEASURES:

1. Primary Outcome: Bone Mineral Density (BMD) at Lumbar Spine (L1-L4)
Description: Percent changes of bone mineral density at lumbar spine (L1-L4) from baseline to 1-year after treatment will be compared and analysed between 2 groups.
Time Frame: 1 year after treatment
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Original Alendronate (Fosamax) | Generic Alendronate (Bonmax)
Number analyzed (Participants) | 70 | 70
percent | 5.54 (6.39) | 5.39 (4.83)

2. Secondary Outcome: Bone Mineral Density (BMD) at Total Hip
Description: Percent changes of bone mineral density at total hip from baseline to 1-year after treatment will be compared and analysed between 2 groups.
Time Frame: 1 year after treatment
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Original Alendronate (Fosamax) | Generic Alendronate (Bonmax)
Number analyzed (Participants) | 70 | 70
percent | 2.48 (4.56) | 2.52 (3.51)

3. Secondary Outcome: Bone Resorption Markers (Serum CTX)
Description: Percent changes of serum bone markers (serum CTX) from baseline to 1-year after treatment will be compared and analysed between 2 groups.
Time Frame: 1 year after treatment
Reporting Status: Not Posted, anticipated posting 2022-04

4. Secondary Outcome: Bone Formation Marker (Serum PINP)
Time Frame: 1 year after treatment
Reporting Status: Not Posted, anticipated posting 2022-04

ADVERSE EVENTS:
Arm/Group | Original Alendronate (Fosamax) | Generic Alendronate (Bonmax)
Serious Adverse Events (participants affected / at risk) | 1/70 | 2/70
Other Adverse Events (participants affected / at risk) | 16/70 | 10/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Original Alendronate (Fosamax) (N=70) | Generic Alendronate (Bonmax) (N=70)
hip fracture (Musculoskeletal and connective tissue disorders) | 1 (70) | 2 (70)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Original Alendronate (Fosamax) (N=70) | Generic Alendronate (Bonmax) (N=70)
myalgia and arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 10

LIMITATIONS AND CAVEATS:
small sample sizes and only one generic brand of bisphosphonate was used.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No